CLINICAL TRIAL: NCT04639791
Title: To Assess the Management of Patients on Global Initiative of Asthma (GINA) Step 4 and 5 Treatment in Hong Kong
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fanny W.S. Ko, Honorary Associate Professor, Chinese University of Hong Kong
Other Study IDs: Severe Asthma Management_v2
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe asthma patients: on step 4& 5 of GINA treatment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observation only, no intervention

SUMMARY:
This study aims to prospectively assess the asthma control and management of asthma patients who are on step 4, 5 asthma of GINA in Hong Kong (on at least medium-dose ICS-LABA as controller therapy for asthma) and also observe their exacerbations over 2 years. In addition, this study will also assess patients who are on biologics for their suitability and outcome. The investigators hope this study will be able to provided data regarding the management and outcome of patients who have difficult-to-treat and severe asthma. The investigators plan to build a biologic registry for asthma that would be able to help local doctors to gain experience to the use of these new and expensive medications.

This is a multi-centre study involving public hospitals in Hong Kong.

This study is important as this will generate local data for healthcare planning for severe asthma in Hong Kong.

DETAILED DESCRIPTION:
Background Asthma is a heterogeneous disease, usually characterized by chronic airway inflammation. It is defined by the history of respiratory symptoms such as wheeze, shortness of breath, chest tightness and cough that vary over time and in intensity, together with variable expiratory airflow limitation.1 The World Health Organization estimates that 300 million people worldwide have asthma with an associated 250,000 asthma deaths annually.2 In Hong Kong, the prevalence rates of physician-diagnosed asthma in 13- to-14-year-olds were 10.2% in 2002,3 and 5.8% in the elderly (aged >70 years) in 2003.4 The crude mortality rate of asthma in 2005 in Hong Kong was 1.4/100,000.5

Severe asthma is not very common but casts a considerable burden on the healthcare system and patients. According to a Dutch survey which included adult asthma patients, 17.4% and 3.6% of them had difficult-to-treat asthma and severe asthma respectively.6 Although severe asthma involves only a small proportion of the asthma population, it generates a huge amount of asthma-related healthcare expenditure.7 An observational cohort by a French study group found that 83% of patients with severe asthma experienced at least one exacerbation and 14% were hospitalised for asthma over the past 12 months.8 Also, patients with severe asthma experience a different spectrum and more severe symptoms, with higher functional and psychological limitation than the general asthma population.9

Asthma is considered as difficult-to-treat if it remains uncontrolled despite Global Initiative for Asthma (GINA) step 4 or 5 treatment (e.g. medium or high dose inhaled corticosteroids [ICS] plus a second controller), or that requires such treatment to maintain good symptom control and reduce the risk of exacerbation.1 Various modifiable factors may contribute to difficult-to-treat asthma, that includes incorrect inhaler technique, suboptimal medication adherence, associated comorbid conditions and even wrong diagnosis. Severe asthma is considered as a subset of difficult-to-treat asthma after exclusion of the modifiable factors other than poorly controlled asthma itself. It is defined as asthma that is uncontrolled despite adherence with maximal optimised therapy and treatment of contributory factors, or that worsens when high dose treatment is decreased.1 Disease phenotyping has revolutionised the management of asthma from stepwise treatment to phenotype-based treatment. As asthma is a clinical syndrome comprising of several spectrums of symptom, different molecular pathways may be involved. Most of these are associated with evidence of cellular inflammation in the airway.10 Identifying treatable traits may potentially guide the choice and predict the outcome of treatment, e.g. blood or airway eosinophilia, is usually a good indicator of corticosteroid responsiveness.11 12 The process of characterising observable treatable traits is termed phenotyping, and this allows physicians to select the most appropriate add-on therapies for patients with severe asthma. Phenotype identification is usually performed in patients on high dose ICS, as most clinical trials on an add-on or biologic treatments were performed in this group of patients.

Among the various inflammatory phenotypes, Type 2 inflammation is the most important one, and its mechanism forms the basis of several biologic treatments. This inflammation pathway is characterised by the presence of interleukin (IL)-4, IL-5 and IL-13. IL-4 and IL-5 promote the production of immunoglobulin E (IgE) and eosinophils respectively, thus the occurrence of eosinophilic inflammation and atopic phenomenon in asthma.1, 13

Five biologics have been approved by the US Food and Drug Administration (FDA) for antagonising the Type 2 inflammatory mechanisms in severe asthma. They are omalizumab, mepolizumab, reslizumab, benralizumab, and dupilumab. In general, severe asthma patients with clinical and laboratory features manifesting Type 2 inflammation (e.g. allergen-driven, high IgE level, high eosinophil activity) and exacerbations are good candidates for such treatment.

In Hong Kong, there is no information regarding the prevalence of severe or difficult to treat asthma. There is also a lack of data on how this group of severe patients are managed, and also their morbidity and mortality. Biologics have been introduced into Hong Kong, and there is no data on how the patients are responding to these new therapies.

Aims of the study This study aims to prospectively assess the asthma control and management of asthma patients who are on step 4, 5 asthma of GINA1 in Hong Kong (on at least medium-dose ICS-LABA as controller therapy for asthma) and also observe their exacerbations over 2 years. In addition, this study will also assess patients who are on biologics for their suitability and outcome. The investigators hope this study will be able to provided data regarding the management and outcome of patients who have difficult-to-treat and severe asthma. The investigators plan to build a biologic registry for asthma that would be able to help local doctors to gain experience to the use of these new and expensive medications.

This is a multi-centre study involving public hospitals in Hong Kong. At the moment, Prince of Wales Hospital and Queen Elizabeth Hospital will join the study. The investigators will invite more hospitals to join later and will get ethical approval in all involved centres.

This study is important as this will generate local data for healthcare planning for severe asthma in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Asthma patients with age ≥18. Asthma is defined as those with a consistent history and prior documented evidence of variable airflow obstruction.
* Subjects on steps 4 and 5 of GINA asthma therapy

Exclusion Criteria:

* Patients with respiratory diseases with other known respiratory diseases including chronic obstructive pulmonary disease, bronchiectasis, tuberculosis (TB)-destroyed lung parenchyma, history of lung resection and lung cancer
* Individuals older than 40 years with a smoking history of more than 10 pack-years
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma patients who are on Steps 4 and 5 of GINA asthma therapy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Level of asthma control | 24 months
  By GINA 2020 criteria of well-controlled, partly controlled or uncontrolled asthma
Asthma Exacerbation | 24 months
  Exacerbation that requires treatment with oral steroid (for patients on maintenance oral steroid, then increase in dose of the oral steroid).
Hospitalization for asthma | 24 months
  Number of hospitalization for asthma

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
No planning yet. Can be shared with no personal data identification to collaborators if needed.